CLINICAL TRIAL: NCT01979367
Title: To Evaluate the Efficacy Treatment of Lower Extremity Pathologies Derived From Neurological Ischemia Disorders
Brief Title: Physician Clinical Trial Policy (CTP) Neurological Ischemia Lower Extremity Pain and Swelling
Acronym: DTSC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Association of Sensory Electrodiagnostic Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTSC030113
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Lower Extremity Swelling Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Anodyne (Experimental): To evaluate the efficacy treatment of lower extremity pathologies from neurological ischemia disorders using the Monochromatic Infrared Photo Energy (MIRE)
  Interventions: Device: Anodyne

INTERVENTIONS:
Device: Anodyne — Subjects will be treated with MIRE therapy using the Anodyne® device within 72 hours of previous treatments, and in accordance with the Anodyne® package insert indications for use 30 to 45 minutes professional units on power setting of 8,. In addition, patients will undergo TENS therapy with the use of either the Avazzia® Pro Sport or TENS 3000 (for no less than 30 mins, both on label) in accordance with the indications for use of each TENS device, for a minimum of 15 minutes at the subjective site for pain and each vertebrae nerve base, when impairment is confirmed with the objective Small Pain Fiber (SPF) Nerve Conduction Study (NCS) test performed.

SUMMARY:
Physician Clinical Trial Policy (CTP) to evaluate the efficacy treatment of lower extremity pathologies derived from neurological ischemia disorders using the combination of Monochromatic Infrared Photo Energy (MIRE) and Transcutaneous Electrical Nerve Stimulation (TENS) therapies.

DETAILED DESCRIPTION:
Although there are a number of pain disorders, associated with back, or lower extremity pain and swelling, the American Association of Sensory Electrodiagnostic Medicine (AASEM/ DTSC) study programs will accumulate received data following a protocol of treatment performed for the purpose of eliminating pain, reducing swelling, and accelerating recovery periods as well as to record the success or failure and/or improvement of the malfunctioning body part.

* Condition: Neuropathic Pain, Tingling or Numbness derived from neurological Ischemia
* Intervention: Treatments of Monochromatic Infrared Photo Energy (MIRE) in combination with Electronic Signal Treatment (TENS) therapy
* Study Type: Interventional
* Study Design:

  1. Allocation: Non-Randomized
  2. Endpoint Classification: Efficacy Study
  3. Intervention Model: Single Group Assignment
  4. Masking: Open Label
  5. Primary Purpose: Scientific record of treatment success or failure

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's judgment, a high probability of 5 year survival and compliance with the study visit schedule.

Ability to comprehend and sign an informed consent document prior to study enrollment.

Exclusion Criteria:

* Any other excluding factors that, according to the investigator's judgment, would preclude enrollment in the study.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-03; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Scientific record of treatment success or failure | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyer, M.D., Study Director — American Association of Sensory Electrodiagnostic Medicine; Chad Pfefer, M.D., Study Chair — American Association of Sensory Electrodiagnostic Medicine

IPD SHARING:
Plan to Share IPD: No